CLINICAL TRIAL: NCT01891240
Title: Personalized Medicine for Pregnant Women: Novel Metabolomic and Proteomic Biomarkers to Detect Pre-eclampsia and Improve Outcome.
Brief Title: IMproved PRegnancy Outcome by Early Detection
Acronym: IMPROvED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Louise Kenny (Other)
Collaborators: Keele University (Other); University of Liverpool (Other); Karolinska University (Other); Erasmus Medical Center (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); MedSciNet AB, Stockholm, Sweden (Unknown); MyCartis, Ghent, Belgium (Unknown); Metabolomic Diagnostics Ltd, Cork, Ireland (Unknown); Accelopment AG (Other); University of Groningen, The Netherlands (Unknown); INFANT centre, University College Cork, Republic of Ireland (Unknown)
Responsible Party: Sponsor-Investigator, Louise Kenny, Professor, University College Cork
Organization: University College Cork (Other)
Other Study IDs: Study Protocol v. 8.0 20122013; Project no: 305169 (Other Grant/Funding Number: FP7-HEALTH-2012-Innovation-1)
Record Dates: First submitted 2013-05-20; First posted 2013-07-03 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Pre-eclampsia; Pregnancy; Pregnancy, High-risk; Pregnancy Complications
Keywords: Diagnostic; Pre-eclampsia; Pregnancy outcome; Mass screening; Diagnostic Techniques and Procedures
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA plasma and serum. Optional urine, hair and baby cord samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- First time, low risk mothers: The study population will consist of first time, low risk mothers attending for antenatal care in one of the participating clinical centres.

SUMMARY:
The overall objective of the IMPROvED project is to develop a sensitive, specific, high-throughput and economically viable early pregnancy screening test for preeclampsia.

This will involve a multicentre, phase IIa clinical predictive study to assess and refine novel and innovative prototype tests based on emerging metabolomic and proteomic technologies developed by SMEs (small to medium size enterprise) within the consortium. The study will i) recruit 5000 first-time pregnant women; ii) establish a high calibre biobank, augmented by accurate clinical metadata; iii) determine whether prototype predictive assays and algorithms translate to the clinical environment; iv) assess potential synergy of a combined metabolomic and proteomic approach and v) progress regulatory approval and development of the selected test into the clinical arena.

DETAILED DESCRIPTION:
Sample size calculations have been considered extensively and given the complexity of the study; there is no single simple solution. For the purpose of sample size estimation in the overall study, we used a binary outcome and associated measures of sensitivity and likelihood ratio as determinants of the value of these tests. Although the predictive algorithms will produce a continuous risk score, the use of a categorical outcome fits with the final binary decision process (to treat or not to treat) based on the risk score. Based on the lowest estimated prevalence of pre-eclampsia of 3% and a test sensitivity of 93% and a test specificity of 97%, then to be 90% certain that the true specificity of the patient population is no less than 95%, a sample size of 4,800 participants is required. Thus, allowing for patient dropout, a study population of 5,000 women is needed.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous.
* Singleton pregnancy, between 9+0 and 16+6 weeks' gestation.
* Signed informed consent.

Exclusion Criteria:

* Unsure of last menstrual period (LMP) and unwilling to have ultrasonography screening (USS) at ≤ 20 weeks.
* ≥ 3 miscarriages.
* ≥3 terminations of pregnancy.
* Known or suspected major fetal anomaly/abnormal karyotype.
* Essential hypertension treated pre-pregnancy.
* Moderate-severe hypertension at booking (BP >160/100 mmHg).
* Diabetes mellitus.
* Renal disease.
* Systemic lupus erythematosus.
* Anti-phospholipid syndrome.
* Sickle cell disease.
* HIV positive.
* Hepatitis B or C positive.
* Major uterine anomaly.
* Cervical suture in situ.
* Knife cone biopsy.
* Long-term steroids.
* Treatment with low-dose aspirin.
* Treatment with heparin/LMW heparin.
* Lack of informed consent.

After recruitment, if the woman is found to be outside the stated gestation limits for the IMPROvED 1st visit of 9 weeks 0 days to 13 weeks 6 days she will be retained in the study if she is willing to take part in the second and third visit and is otherwise eligible. There is one pre-specified criteria for discontinuation of a participant. If a woman is recruited into the IMPROvED study and later identified as having a pregnancy exclusion criterion, i.e., ≥ 3 miscarriages, ≥ 3 TOPS, or using low-dose aspirin at the time of recruitment, she shall be excluded. However, women diagnosed during the pregnancy but after recruitment with an exclusion criterion, e.g., diseases such as renal disease, anti-phospholipid syndrome, etc. shall be retained within the study. Women who are recruited but later discontinue from the study do not count towards recruitment targets for each centre. Accordingly, such dropouts must be replaced.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: First time, low risk mothers attending antenatal care units. Women will be referred to IMPROvED through a number of routes including referral by their midwife, obstetrician or general practitioner and self-referral following exposure to the study through friends, posters, advertisements, website and news stories. Maternity caregivers in each centre will provide information about the study to eligible women in early pregnancy.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-10 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Pre-eclampsia. | 7 days after birth
  Preeclampsia is defined as gestational hypertension defined as systolic BP ≥140mmHg and/or diastolic BP ≥90mmHg (Korotkoff V) on at least 2 occasions 4h apart after 20 weeks' gestation, but before the onset of labour or postpartum systolic BP ≥140mmHg and/or diastolic BP ≥90mmHg on at least 2 occasions 4h apart with either proteinuria ≥300mg/24h or spot urine protein:creatinine ratio ≥30mg/mmol creatinine or urine dipstick protein ≥++.
Spontaneous pre-term birth | Up to 37+0 weeks´ gestation
  Spontaneous pre-term birth is defined as spontaneous preterm labour or preterm premature rupture of the membranes resulting in preterm birth at <37+0 weeks' gestation.
Small for gestational age (SGA) | Within 24 hours after birth
  The birth weight is converted to a customized centile, adjusting for gestation, maternal weight, height, parity, ethnicity and infant sex. SGA is defined as <10th customised centile.

SECONDARY OUTCOMES:
Early onset pre-eclampsia | Followed for the duration of hospital stay, an expected average of 6 weeks
  Pre-eclampsia resulting in delivery at <34+0 weeks' gestation.
Multisystem complications of pre-eclampsia | Between 20 weeks´gestation and 6 weeks after birth
  Defined as one or more of the following:
  * Acute renal insufficiency defined as new increase in serum creatinine to >100μmol/L antepartum or >130μmol/L postpartum.
  * Liver disease defined as raised aspartate transaminase and/or alanine transaminase >45 IU/L and/or severe right upper quadrant or epigastric pain or liver rupture.
  * Neurological problems defined as eclampsia, imminent eclampsia (severe headache with hyperreflexia and persistent visual disturbance) or cerebral haemorrhage.
  * Haematological abnormalities including thrombocytopenia (platelets <100x109/L), disseminated intravascular coagulation or haemolysis, diagnosed by features on blood film (such as fragmented cells, helmet cells) and reduced haptoglobin.
Pre-eclampsia with severe fetal or neonatal complications | Followed for the duration of hospital stay, an expected average of 6 weeks
  Pre-eclampsia resulting in either delivery at < 32+0 weeks' gestation or major neonatal morbidity or stillbirth or neonatal death or post-neonatal death.
Major neonatal morbidity in preterm infants | Followed for the duration of hospital stay, an expected average of 6 weeks
  One or more of the following amongst babies delivered before 37 weeks' gestation:
  Grade III or IV intraventricular haemorrhage; Chronic lung disease; Necrotizing enterocolitis; Retinopathy of prematurity stage 3 or 4; Sepsis (blood or CSF culture proven); Or cystic periventricular leukomalacia. These conditions will be defined using the Australian and New Zealand neonatal network definitions.
Major neonatal morbidity in term infants | Followed for the duration of hospital stay, an expected average of 6 weeks
  One or more of the following amongst babies delivered at or after 37 weeks' gestation:
  Grade II or III hypoxic ischaemic encephalopathy; Ventilation >24 hours; Neonatal unit care admission >4 days; Apgars < 4 at 5 minutes; Cord arterial pH <7.0 and/or base excess >-15; Or neonatal seizures.
Pre-eclampsia with severe maternal complications | Followed for the duration of hospital stay, an expected average of 6 weeks
  The development of pre-eclampsia with one or more of the following:
  Maternal death; Persistent severe hypertension (systolic blood pressure ≥170mmHg or diastolic blood pressure ≥110mmHg on more than one occasion antepartum or postpartum); Or multi-system complication (as defined in outcome above.
Preeclampsia with either severe maternal complication or severe fetal or neonatal complications | Followed for the duration of hospital stay, an expected average of 6 weeks
  Pregnancies affected by severe maternal or severe fetal or neonatal complications (as defined in Major neonatal morbidity in preterm infants or Major neonatal morbidity term infants).
Early onset SGA | Followed for the duration of hospital stay, an expected average of 6 weeks
  SGA resulting in delivery at <34+0 weeks' gestation.
SGA with severe fetal or neonatal complications | Followed for the duration of hospital stay, an expected average of 6 weeks
  SGA and either delivery at <32+0 weeks' gestation or major neonatal morbidity (as defined in Major neonatal morbidity in preterm infants) or stillbirth or neonatal death or post-neonatal death.
Early onset spontaneous preterm birth | Followed for the duration of hospital stay, an expected average of 6 weeks
  Spontaneous pre-term birth resulting in delivery < 34+0 weeks' gestation.
Spontaneous preterm birth with severe fetal or neonatal complications | Followed for the duration of hospital stay, an expected average of 6 weeks
  Spontaneous preterm birth (PTB) resulting in either delivery at <32+0 weeks' or spontaneous PTB resulting in major neonatal morbidity (as defined in Major neonatal morbidity in preterm infants) or stillbirth or neonatal death or post-neonatal death.
Spontaneous preterm birth with PPROM | Followed for the duration of hospital stay, an expected average of 6 weeks
  Spontaneous PTB following preterm premature rupture of the membranes (PPROM).
Spontaneous preterm birth without PPROM | Followed for the duration of hospital stay, an expected average of 6 weeks
  Spontaneous PTB with intact membranes at the onset of labour.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Kenny, Professor, Principal Investigator — INFANT Centre, University College Cork, Ireland; Philip N Baker, Professor, Principal Investigator — Keele Univeristy School of Medicine
Locations (6):
- Cork University Maternity Hospital, University College Cork, Wilton, Cork, Ireland
- Erasmus Medical Center Rotterdam, Rotterdam, Netherlands
- Karolinska University Hospital Huddinge, Karolinska Institute, Stockholm, Sweden
- United Kingdom (3):
  - Liverpool Women's Hospital, University of Liverpool, Liverpool, Merseyside
  - Keele University School of Medicine, Shrewsbury and Telford Hospital NHS Trust, Shrewsbury, Shropshire
  - Keele University School of Medicine, University Hospital of North Midlands, Stoke-on-Trent, Staffordshire

REFERENCES:
- [Derived] McCarthy EK, Schneck D, Basu S, Xenopoulos-Oddsson A, McCarthy FP, Murray DM, Georgieff MK, Kiely ME. Impact of Maternal Iron Deficiency in Early Pregnancy on Neonatal Iron Status and Neurodevelopment at Two Years of Age: a Prospective, Maternal-Infant Cohort Study. J Nutr. 2026 Jan;156(1):101240. doi: 10.1016/j.tjnut.2025.11.009. Epub 2025 Nov 12. PMID 41238120
- [Derived] McCarthy EK, Schneck D, Basu S, Xenopoulos-Oddsson A, McCarthy FP, Kiely ME, Georgieff MK. Longitudinal evaluation of iron status during pregnancy: a prospective cohort study in a high-resource setting. Am J Clin Nutr. 2024 Nov;120(5):1259-1268. doi: 10.1016/j.ajcnut.2024.08.010. Epub 2024 Sep 26. PMID 39510727
- [Derived] Navaratnam K, Alfirevic Z, Baker PN, Gluud C, Gruttner B, Kublickiene K, Zeeman G, Kenny LC. A multi-centre phase IIa clinical study of predictive testing for preeclampsia: improved pregnancy outcomes via early detection (IMPROvED). BMC Pregnancy Childbirth. 2013 Dec 7;13:226. doi: 10.1186/1471-2393-13-226. PMID 24314209
- See also: Official website of IMPROvED — http://www.fp7-improved.eu/